CLINICAL TRIAL: NCT04528914
Title: Effect of a Low-FODMAP Diet for the Management of Functional Abdominal Pain Disorders in Children
Brief Title: Low-FODMAP Diet for Functional Abdominal Pain Disorders in Children.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary results found that there is no difference on abdominal pain intensity between low-FODMAP and regular diet at 4 weeks. Moreover, both diets were difficult to adhere by patients. We do not expect any significant change in our findings.
Sponsor: Medical University of Warsaw (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1W44/5FNUT13/20
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-02

CONDITIONS: Functional Abdominal Pain Disorder
Keywords: functional abdominal pain disorders; irritable bowel syndrome; diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research investigators, outcome assessor, and independent statistician (data analyst) will be blinded until the completion of the data analysis.The dietitian will remain unblinded. Success of blinding will be assessed after completion of the follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-FODMAP diet (Experimental): 37 participants.
  Interventions: Other: Low-FODMAP diet
- Regular diet (No Intervention): 37 participants. The regular diet will reflect the habitual FODMAP intake in a normal diet.
  Diets in both groups will be matched in terms of total energy, fat, protein, carbohydrates and dietary fiber with the usual participant's diet.

INTERVENTIONS:
Other: Low-FODMAP diet — The low-FODMAP diet will contain the amount of FODMAPs that will not exceed the cut-offs for each FODMAP sugar per serving of food per sitting. Diets will be individually tailored by dietitian and delivered by a catering company (five meals each day).
  Arms: Low-FODMAP diet

SUMMARY:
This single-center, randomized, controlled, quadruple-blinded, superiority trial is performed to test the hypothesis that children with IBS and FAP-NOS who receive a low-FODMAP diet will have a lower mean abdominal pain intensity score compared with those who receive a regular diet after 4 weeks of intervention.

DETAILED DESCRIPTION:
Introduction. Evidence from studies in adults documents that fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAPs) may be triggers of symptoms in individuals with functional abdominal pain disorders. However, in children with FAPDs, there is a need for high-quality evidence regarding the dietary management. We aim to assess the effects of a low-FODMAP diet compared with a regular diet for the management of children with FAPDs.

Methods. In this trial, seventy-four children aged 8 to 18 years with a Functional Abdominal Pain Disorder (Irritable Bowel Syndrome or Functional Abdominal Pain-Not Otherwise Specified), diagnosed according to the Rome IV criteria, will be randomly allocated to receive either a low-FODMAP diet or a regular diet for 4 weeks.A primary outcome will be the percentage of the responders, defined as the participants who have at least 30% improvement in abdominal pain intensity on a Visual Analogue Scale (VAS) during the last week of the trial compared with baseline, that is at least equal to the Reliable Change Index (≥ 25 mm change on VAS).

ELIGIBILITY:
Inclusion Criteria:

* functional abdominal pain - not otherwise specified (FAP-NOS) or irritable bowel syndrome (IBS) diagnosed according to the Rome IV Criteria,
* baseline average pain intensity at least 30 mm on a 100-mm Visual Analogue Scale,
* feeding via the oral route,
* ability to read and comprehend any employed questionnaires/scales,
* signed informed consent,
* stated availability throughout the study period.

Exclusion Criteria:

* receiving any other intervention/treatment with regard to FAP-NOS or IBS or those who received any other intervention during the last 3 months,
* an organic cause of symptoms or organic gastrointestinal disease,
* chronic illness, receiving medications which affect gastrointestinal motility,
* need for any other dietary management which could make the balancing or compliance with the diet troublesome,
* previously diagnosed carbohydrate intolerance without symptoms of FAPD after implementation of an exclusion diet,
* undernutrition (defined as World Health Organization [WHO] growth charts < -2 SD), decreased growth velocity (sharp decline in growth line), or overweight or obese (> 1 or > 2 SD on the WHO growth charts, respectively),
* unintentional weight loss greater or equal to 5% of subject' body weight within the previous 3 months,
* pregnancy,
* eating disorders,
* prior surgery of the gastrointestinal tract (within last 3 months),
* recurrent or unexplained fever,
* developmental disabilities which impair the ability of the child to understand or communicate.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in abdominal pain intensity | At week 1, 2, 3 and 4 from baseline.
  The primary outcome will be the percentage of the responders, defined as the participants who have at least 30% improvement in abdominal pain intensity on a 100-mm Visual Analogue Scale (VAS) during the last week of the trial compared with baseline, that is at least equal to the Reliable Change Index (≥ 25 mm change on VAS).

SECONDARY OUTCOMES:
Change in stool consistency | At week 1, 2, 3 and 4 from baseline.
  Bristol Stool Scale is a seven-point scale that distinguish seven pictures of different forms of stool, ranging from the hardest (type 1) to the softest (type 7).
  At baseline, participants with IBS and a stool consistency score > 5 on the Bristol Stool Scale will be classified as having IBS with predominant diarrhea (IBS-D); if the stool consistency score is < 3, the subjects will be classified as having IBS with predominant constipation (IBS-C).
  Responders will be subjects with improvement in their average stool consistency during the last week of the trial compared with baseline [≥1 higher Bristol Stool Scale score in case of IBS with predominant constipation, or at least one lower score in case of IBS with predominant diarrhea].
Change in abdominal pain frequency | At week 1, 2, 3 and 4 from baseline.
Change in Gastrointestinal Symptom Rating Scale (GSRS) total score | At week 1, 2, 3 and 4 from baseline.
  The GSRS is a 15-item interview-based rating scale. Each item is assessed in a seven-point graded Likert-type scale (one means no symptoms, and seven represents very troublesome symptoms), then total score is calculated.
Change in KIDSCREEN-10 index total score | At week 1, 2, 3 and 4 from baseline.
  KIDSCREEN-10 index is a 11-item instrument to assess health-related quality of life (HRQoL). Each item is assessed in a 5-point scale with higher values indicating a higher HRQoL. Total score is calculated.
Change in World Health Organization Five Well-Being Index (WHO-5) total score | At week 1, 2, 3 and 4 from baseline.
  The WHO-5 consists of five statements regarding the physical well-being, assessed in a six-point scale (in which zero means at no time, and five represents all of the time). Total raw score is then calculated, ranging from 0 to 25 which is multiplied by four, therefore the final score ranges from 0 (the worst imaginable well-being) to 100 (the best imaginable well-being).
Change in percentage of school attendance associated with IBS symptoms | At week 1, 2, 3 and 4 from baseline.
Change in percentage of parents' work absenteeism associated with IBS symptoms in child | At week 1, 2, 3 and 4 from baseline.
Change in BMI-for-age z-score | At week 2 and 4 from baseline.
  The body weight (kg) and standing height (cm) will be measured following standard methods. Body Mass Index (BMI) will be calculated using the standard equation. BMI-for-age z-score will be computed using the WHO AnthroPlus software v1.0.4., then assessed and monitored over time using the WHO growth charts.
Percentage of compliant participants | 0-4 weeks.
  The percentage compliance in each group will be calculated. A compliant participant is considered as one who consumes at least 80% of the provided diet.
  The percent of each meal which the subject consumed (<50%, 50-79% or 80-100%) each day will be reported by participant in a study diary (developed by research team); the additional snacks consumed also will be reported daily (characteristics and amount). Snacks and meals outside the meal plan will be assessed separately.
Percentage of tolerability of the low-FODMAP diet | 0-4 weeks.
  The tolerability (acceptability) of the diet will be assessed each day using a 100-mm Visual Analogue Scale and reported in the subject diary. This outcome will be reported as a mean for each study group, and as a comparison between groups.
Adverse events | 0-4 weeks.
  The number of all adverse events and the number of participants reporting adverse events associated with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or generated during this study will be made available after the publication of results, no later than 3 years from the completion of data analysis.
Supporting Information: CSR
Time Frame: Up to 3 years after completion of data analysis.
Access Criteria: The datasets will be made available from the contact author upon reasonable request.

REFERENCES:
- [Derived] Strozyk A, Horvath A, Muir J, Szajewska H. Effect of a low-FODMAP diet for the management of functional abdominal pain disorders in children: a study protocol for a randomized controlled trial. Nutr J. 2021 Jan 2;20(1):1. doi: 10.1186/s12937-020-00656-3. PMID 33388067